CLINICAL TRIAL: NCT00928460
Title: The Efficacy of Routine Preoperative Electrocardiography in Patients Undergoing Non-cardiac Surgery
Brief Title: Efficacy of Preoperative Electrocardiography
Status: Withdrawn | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Wilton A van Klei, MD PhD, UMC Utrecht
Other Study IDs: ECGtrial
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Cardiac Arrest
Keywords: Electrocardiogram; Electrocardiography; Perioperative care; Preoperative care; Preanesthesia Evaluation; Acute Coronary Syndrome; Postoperative Myocardial Infarction; Myocardial ischaemia; Postoperative Cardiac Death; Intraoperative complications; Postoperative complications; Cost-effectiveness analysis
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Heart Arrest; Coronary Artery Disease; Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Regular preanesthesia evaluation: Patients are evaluated by the anesthesiologist according to current protocol, including routine preoperative ECG.
- New preanesthesia evaluation: Patients are evaluated by the anesthesiologist according to a new protocol, in which a routine preoperative ECG is no longer provided.
  Interventions: Procedure: Removal of preoperative electrocardiogram

INTERVENTIONS:
Procedure: Removal of preoperative electrocardiogram — A new preanesthesia evaluation strategy without routine ECG. Initially, all patients in the participating centers are assessed following the regular strategy (with routine ECG). The new strategy (without routine ECG) is rolled out to the participating hospitals sequentially. At the end of the trial all participating centers will use the new preoperative strategy.
  Groups: New preanesthesia evaluation

SUMMARY:
A preoperative electrocardiogram (ECG) is nearly routinely performed by anesthesiologists in elderly non-cardiac surgery patients as part of pre-anesthesia evaluation. However, the added value of this routine ECG beyond patient history and physical examination is questionable. The ECGtrial will investigate the efficacy of routine preoperative electrocardiography in patients undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Objective:

A routine ECG is performed as part of the standard diagnostic workup before non-cardiac surgery. However, the added value of this test beyond patient history and physical examination is questionable. The proposed study therefore aims to determine whether preoperative assessment without ECG is more cost-effective.

Study design:

Prospective stepped wedge design multicenter trial including 40,000 patients.

Study population:

All patients aged over 60 years, or younger patients with cardiovascular risk factors, scheduled for non-cardiac surgery with an expected postoperative hospital stay of at least 2 days.

Intervention:

A new preoperative assessment strategy without routine ECG. Initially, all patients in the participating centers are assessed following the regular strategy (with routine ECG). The new strategy (without routine ECG) is rolled out to the participating hospitals sequentially. At the end of the trial all participating centers will use the new preoperative strategy.

Outcome measures:

The primary outcome measure is cardiac death or perioperative myocardial infarction. The latter will be verified by Troponin values at postoperative day 1 and 2. If the Troponin levels are elevated the presence of myocardial infarction will be evaluated by a consulting cardiologist. Secondary outcomes are other major cardiovascular complications, death from other causes within 2 days of surgery, and long term quality of life. To determine cost-effectiveness of the strategy without ECG all pre- and postoperative referrals and interventions are taken into account.

Sample size calculation:

We expect no increase in the primary outcome in the intervention group. To rule out an 0.5% increase (from 3% to 3.5%) in the intervention group, the inclusion of 36,504 patients is required (level of confidence: 0.95; power: 0.80). To compensate for expected 10% loss-to-follow up, 40,000 patients will be randomized.

Economic evaluation:

A cost-effectiveness analysis will be conducted when the increase in primary outcome is between 0.0 and 0.5%. If the intervention results in a lower prevalence of the primary outcome, no cost-effectiveness analysis is performed as the health and cost outcomes point in the same, advantageous, direction. An increase of more than 0.5% is not considered acceptable from a clinical point of view.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 60 years or older scheduled for noncardiac surgery with an expected hospital length of stay of at least 2 days
* Patients aged under 60 years but with risk factors for cardiovascular disease scheduled for noncardiac surgery with an expected hospital length of stay of at least 2 days

Exclusion Criteria:

* Patients refusing informed consent for obtaining blood samples (troponin measurement) at the first two days after surgery
* Patients refusing participation in long-term clinical and Quality of Life measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged over 60 years, or younger patients with cardiovascular risk factors, scheduled for non-cardiac surgery with an expected postoperative hospital length of stay of at least 2 days.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Cardiac death or perioperative myocardial infarction | 2 days postoperatively

SECONDARY OUTCOMES:
Other major cardiovascular complications | 2 days postoperatively
Death from other causes | 2 days postoperatively
Long term quality of life | One year

CONTACTS AND LOCATIONS:
Overall Officials: Cor J Kalkman, MD PhD, Study Chair — UMC Utrecht; Wilton A van Klei, MD PhD, Principal Investigator — UMC Utrecht; Jurgen C de Graaff, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] van Klei WA, Bryson GL, Yang H, Kalkman CJ, Wells GA, Beattie WS. The value of routine preoperative electrocardiography in predicting myocardial infarction after noncardiac surgery. Ann Surg. 2007 Aug;246(2):165-70. doi: 10.1097/01.sla.0000261737.62514.63. PMID 17667491